CLINICAL TRIAL: NCT03586128
Title: Integrated PrEP and ART Delivered in Ugandan Public Health Clinics to Improve HIV and ART Outcomes for HIV Serodiscordant Couples
Brief Title: Partners PrEP Program
Acronym: PPP
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: Harvard University (Other); Makerere University (Other)
Responsible Party: Principal Investigator, Renee Heffron, Assistant Professor, School of Public Health: Global Health, University of Washington
Other Study IDs: STUDY00000320
Record Dates: First submitted 2018-06-19; First posted 2018-07-13 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HIV serodiscordant couples
  Interventions: Drug: PrEP; Drug: ART

INTERVENTIONS:
Drug: PrEP — PrEP will be introduced into clinics according to Uganda national guidelines using a stepped wedge design. Uganda guidelines recommend any tenofovir disoproxil fumarate (TDF) containing medication be used for PrEP; this includes emtricitabine (FTC)/TDF, lamivudine (3TC)/TDF or TDF alone.
Drug: ART — ART medication will be provided according to Uganda national guidelines for persons living with HIV.

SUMMARY:
Through close collaboration with the Ugandan Ministry of Health, the investigators plan to provide PrEP for HIV-negative members of HIV serodiscordant couples by launching PrEP delivery within 12 public ART clinics in Kampala, Uganda. Intervention delivery will be launched in a staggered fashion among clinics through a stepped wedge cluster randomized trial providing a rigorous research opportunity to measure the effect of the intervention on PrEP and ART initiation and adherence. To measure these outcomes using clinic records and biomarkers, the program will enroll approximately 1440 HIV serodiscordant couples. Additionally, the program will collect qualitative and quantitative data to determine if PrEP-taking is a modeled behavior that facilitates ART use and characterize the way that PrEP and ART use interact within couples and estimate the programmatic costs of the integrated PrEP and ART strategy.

ELIGIBILITY:
Inclusion Criteria:

For both members of the couple

* Age ≥18 years
* Able and willing to provide informed consent
* Sexually active with each other
* Willing to engage with the clinic system as a couple

For HIV-positive members of the couples (index participants)

* HIV-positive, according to national HIV testing algorithm
* Recent diagnosis as a member in an HIV serodiscordant couple
* Not currently enrolled in an HIV treatment clinical trial

For HIV-negative members of the couples (partner participants)

* HIV-negative, according to national HIV testing algorithm
* Recent diagnosis as a member in an HIV serodiscordant couple
* Not currently enrolled in an HIV treatment clinical trial
* Not currently using PrEP
* Eligible for PrEP, according to WHO or Ugandan national guidelines

Exclusion Criteria:

- Otherwise not eligible based on the above inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV serodiscordant couples from the Kampala, Uganda area
Sampling Method: Non-Probability Sample
Enrollment: 1381 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Number of HIV-positive members of a discordant partnership who initiate ART | Up to 24 months
  Measure ART initiation of the HIV-positive member of the couple
HIV viral load suppression of HIV-positive members of a discordant partnership | Up to 24 months
  ART adherence by measuring HIV viral load of the HIV-positive member of the couple
Number of HIV-negative members of a discordant partnership who initiate PrEP | Up to 24 months
  Measure PrEP initiation of the HIV-negative member of the couple
PrEP adherence of HIV-negative members of a discordant partnership | Up to 24 months
  Measure PrEP adherence, among HIV-negative members of a discordant partnership who initiated PrEP, by self-report and tenofovir drug level testing.

SECONDARY OUTCOMES:
PrEP-taking as a modeled behavior | Up to 24 months
  Measure the degree to which PrEP-taking behavior is modeled by HIV-negative partners and the degree to which it is witnessed by HIV-positive partners using questionnaires developed for this purpose.
Facilitators and barriers to use of ART and PrEP | Up to 24 months
  Mixed methods assessment of how integrated PrEP and ART is 1) used among couples and 2) implemented by health care providers using qualitative interviews and questionnaires. These data will be aggregated to understand the facilitators and barriers to use of ART and PrEP.
Programmatic costs of providing integrated PrEP and ART to HIV serodiscordant couples | Up to 24 months
  Conduct micro-costing, cost-effectiveness, and budget impact analyses to estimate the programmatic costs of providing integrated PrEP and ART to HIV serodiscordant couples.

CONTACTS AND LOCATIONS:
Overall Officials: Renee Heffron, PhD, MPH, Principal Investigator — University of Washington
Locations (1):
- Makerere University, Kampala, Uganda

REFERENCES:
- [Derived] Wyatt MA, Pisarski EE, Nalumansi A, Kasiita V, Kamusiime B, Nalukwago GK, Thomas D, Muwonge TR, Mujugira A, Heffron R, Ware NC; Partners PrEP Program Study Team. How PrEP delivery was integrated into public ART clinics in central Uganda: A qualitative analysis of implementation processes. PLOS Glob Public Health. 2024 Mar 7;4(3):e0002916. doi: 10.1371/journal.pgph.0002916. eCollection 2024. PMID 38452111
- [Derived] Heffron R, Muwonge TR, Thomas KK, Nambi F, Nakabugo L, Kibuuka J, Thomas D, Feutz E, Meisner A, Ware NC, Wyatt MA, Simoni JM, Katz IT, Kadama H, Baeten JM, Mujugira A; Partners PrEP Program Team. PrEP uptake and HIV viral suppression when PrEP is integrated into Ugandan ART clinics for HIV-negative members of HIV-serodifferent couples: A stepped wedge cluster randomized trial. EClinicalMedicine. 2022 Aug 11;52:101611. doi: 10.1016/j.eclinm.2022.101611. eCollection 2022 Oct. PMID 35990584